CLINICAL TRIAL: NCT02342171
Title: Emergency Evaluation of Convalescent Plasma for Ebola Viral Disease (EVD) in Guinea
Acronym: Ebola-Tx
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: National Blood Transfusion Centre (NBTC), Conakry, Guinea (Unknown); Gamal Abdel Nasser University of Conakry (Other); National Center for Training and Research of Maferinyah, Guinea (Unknown); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); University of Oxford (Other); University of Liverpool (Other); London School of Hygiene and Tropical Medicine (Other); Aix Marseille Université (Other); UBIVE, Institut Pasteur, Paris, France (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Etablissement Français du Sang (Other); Belgian Red Cross (Other); Institut Pasteur, Dakar, Sénégal (Unknown); Médecins Sans Frontières, Belgium (Other); World Health Organization (Other); International Severe Acute Respiratory and Emerging Infection Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITM0614
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Ebola Viral Disease; Convalescent Plasma; Developing Countries
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Convalescent Plasma (Experimental): Convalescent Plasma: 400-500 mL from two donors (2 x 200-250 ml) and 10mL/kg for small adults and children <45kg
  Interventions: Other: Convalescent Plasma
- standard care (No Intervention): The control arm will consist of historical controls having being treated with standard of care

INTERVENTIONS:
Other: Convalescent Plasma — Patients will be treated with plasma from recovered EVD patients.
  Arms: Convalescent Plasma

SUMMARY:
This is an emergency, phase 2/3, open-label, non-randomized, clinical trial that will evaluate Convalescent Plasma (CP) added to standardized supportive care (SC) in patients with confirmed Ebola Virus Disease (EVD). No patient will be refused CP when compatible products are available and all efforts will be made to maximize CP availability during the study. EVD patients recruited during the period before CP becomes available or for whom no compatible CP is available will be given SC and will be followed for study outcomes. Data from these SC patients will be the used as comparator in the analysis of the study. The primary objective of the study is to assess if CP + SC improves the 14 day survival of patients, compared to SC alone.

The Investigators aim to enroll a total number of 130 - 200 patients who will be treated treated with CP assuming equal numbers of patients treated with SC alone. If there would be insufficient patients treated with SC, patients treated at the research site prior to study start may be included in the comparison group.

Patients will be recruited in the Ebola Treatment centre managed by Medecins Sans Frontieres (MSF) in Conakry, Guinea. All patients and/or relatives presenting at the centre will be informed about the study, and will be invited to provide consent at the time of admission inside the treatment centre. Only patients for whom ebola infection is confirmed with polymerase chain reaction (PCR) will be enrolled in the study. After inclusion, eligibility to the intervention will be reassessed on regular intervals. If the eligibility criteria are not met by 48 hours after inclusion, only SC will be continued.

In line with the guidance of the World Health Organization (WHO), two units of CP will be given. EVD patients will be transfused with ABO-compatible CP using standard procedures. Details on the modalities of transfusion can be found in the WHO guidance document and the MSF guidelines on blood transfusion. All patients will be under close observation for transfusion-related adverse reactions during and up to 4 hours after transfusion. 24 hours after the start of transfusion, a blood sample will be collected for viral load assessment. All other aspects of patient management will be according to MSF clinical guidelines. The decision to discharge a patient should be taken on clinical grounds, but can be supported by the laboratory results. After discharge, the patient will be followed up by the study team until day 30.

DETAILED DESCRIPTION:
West-Africa is being ravaged by the worst outbreak of Ebola Viral Disease (EVD) ever witnessed. Nine months after its onset, the outbreak has spiraled and currently appears to be out of control. One of the key factors contributing to the high mortality is the lack of any proven effective EVD specific treatment. The identification of effective therapies is a medical and public health priority. Convalescent whole blood (CWB) and convalescent plasma (CP) have been prioritized by the World Health Organization (WHO) to be evaluated within a short time span, so that widespread use for therapy could be implemented rapidly if proven effective. Both CWB and CP contain EBV antibodies and either could potentially be of value as EVD therapy, however their efficacy in Ebola must still be demonstrated. .

This is an emergency, phase 2/3, open-label, non-randomized, clinical trial that will evaluate CP added to standardized supportive care (SC) in patients with confirmed EVD. No patient will be refused CP when compatible products are available and all efforts will be made to maximize CP availability during the study. EVD patients recruited during the period before CP becomes available or for whom no compatible CP is available will be given SC and will be followed for study outcomes. Data from these SC patients will be the used as comparator in the analysis of the study.

The primary objective of the study is to assess if CP + SC improves the 14 day survival of patients, compared to SC alone. Secondary objectives are;

* to assess 30 day survival on CP + SC
* to assess the relationship between EV antibody levels in donated CP and survival in patients receiving CP
* to assess the relationship between EV antibody levels in donated CP and changes in levels of viral RNA in the blood of patients receiving CP
* to assess the occurrence of serious adverse reactions (SARs) related to CP transfusion in Ebola patients
* to assess the occurrence of safety risks related to CP transfusion in health workers administering the treatments
* to determine risk factors for mortality despite administration of CP (for identification of patients most likely to benefit)

The Investigators aim to enroll a total number of 130 - 200 patients treated with CP assuming equal numbers of patients treated with SC alone. The number of patients treated with SC will be determined by the time interval for CP to become available for treatment and the availability of CP throughout the study. If there would be insufficient patients treated with SC, patients treated at the research site prior to study start may be included in the comparison group.

Patients will be recruited in the Ebola Treatment centre managed by Medecins Sans Frontieres (MSF) in Conakry. All patients and/or relatives presenting at the centre will be informed about the study, and will be invited to provide consent at the time of admission inside the treatment centre. Only patients for whom ebola infection is confirmed via polymerase chain reaction (PCR) will be enrolled in the study. After inclusion, eligibility to the intervention will be assessed at the time of enrollment (when the patient is moved to the area for patients with confirmed Ebola) and will be reassessed on regular intervals as long as the patient did not receive plasma transfusion. The re-assessment of eligibility to receive CP happens at 8h and at 12h, and is repeated until 48 hours after inclusion. If the eligibility criteria are not met by 48 hours after inclusion, only SC will be continued.

A patient is not eligible to receive CP if they meet one of the following criteria:

* History of allergic reaction to blood or plasma products (as judged by the investigator or treating physician); (this first criterion is definite and will not be re-assessed)
* Medical conditions in which receipt of additional fluid related to the transfusion (250-500 ml or in the case of children 10 ml/kg) may be detrimental to the patient (e.g. decompensated congestive heart failure or renal failure).
* Patients in shock unresponsive to fluid challenge
* Patients in shock with signs of multi-organ failure, defined as oliguria/anuria AND impaired consciousness AND/OR jaundice
* Condition of patient where the procedure of plasma administration carries a risk for the staff

In line with the WHO guidance, two units of CP will be given. EVD patients will be transfused with ABO-compatible CP using standard procedures. Details on the modalities of transfusion can be found in the WHO guidance document and the MSF guidelines on blood transfusion. All patients will be under close observation for transfusion-related adverse reactions during and up to 4 hours after transfusion. 24 hours after the start of transfusion, a blood sample will be collected for viral load assessment. All other aspects of patient management will be according to MSF clinical guidelines.

The decision to discharge a patient should be taken on clinical grounds, but can be supported by the laboratory results. After discharge, the patient will be followed up by the study team until day 30.

ELIGIBILITY:
Inclusion Criteria:

* PCR-confirmed, symptomatic infection with Ebola virus
* Patient's, guardian's or representatives' willingness to provide written informed consent

Exclusion Criteria:

A patient is not eligible to receive CP if they meet one of the following criteria:

* History of allergic reaction to blood or plasma products (as judged by the investigator or treating physician);
* Medical conditions in which receipt of additional fluid related to the transfusion (250-500 ml or in the case of children 10 ml/kg) may be detrimental to the patient (e.g. decompensated congestive heart failure or renal failure).
* Patients in shock unresponsive to fluid challenge
* Patients in shock with signs of multi-organ failure, defined as oliguria/anuria AND impaired consciousness AND/OR jaundice
* Condition of patient where the procedure of plasma administration carries a risk for the staff

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan van Griensven, MD, Study Chair — ITM; Niankoye Haba, MD, Principal Investigator — National Blood Transfusion Centre (NBTC), Conakry, Guinea
Locations (1):
- Ebola Treatment Center, Donka, Guinea

REFERENCES:
- [Result] van Griensven J, Edwards T, de Lamballerie X, Semple MG, Gallian P, Baize S, Horby PW, Raoul H, Magassouba N, Antierens A, Lomas C, Faye O, Sall AA, Fransen K, Buyze J, Ravinetto R, Tiberghien P, Claeys Y, De Crop M, Lynen L, Bah EI, Smith PG, Delamou A, De Weggheleire A, Haba N; Ebola-Tx Consortium. Evaluation of Convalescent Plasma for Ebola Virus Disease in Guinea. N Engl J Med. 2016 Jan 7;374(1):33-42. doi: 10.1056/NEJMoa1511812. PMID 26735992
- [Result] van Griensven J, Edwards T, Baize S; Ebola-Tx Consortium. Efficacy of Convalescent Plasma in Relation to Dose of Ebola Virus Antibodies. N Engl J Med. 2016 Dec 8;375(23):2307-2309. doi: 10.1056/NEJMc1609116. Epub 2016 Nov 14. No abstract available. PMID 27959686
- [Derived] Edwards T, Semple MG, De Weggheleire A, Claeys Y, De Crop M, Menten J, Ravinetto R, Temmerman S, Lynen L, Bah EI, Smith PG, van Griensven J; Ebola_Tx Consortium. Design and analysis considerations in the Ebola_Tx trial evaluating convalescent plasma in the treatment of Ebola virus disease in Guinea during the 2014-2015 outbreak. Clin Trials. 2016 Feb;13(1):13-21. doi: 10.1177/1740774515621056. Epub 2016 Jan 14. PMID 26768570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convalescent Plasma | Standard Care
Started | 99 | 507
Completed | 84 | 418
Not Completed | 15 | 89
Not completed — Death | 4 | 87
Not completed — Received favipiravir | 10 | 0
Not completed — Missing cycle treshold value | 1 | 0
Not completed — Unknown outcome | 0 | 1
Not completed — Missing age data | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Plasma | Standard Care | Total
Number analyzed (Participants) | 84 | 418 | 502
Age, Continuous [Median (Full Range); unit: years] | 29 [0 to 75] | 28 [0 to 87] | 28 [0 to 87]
Age, Customized [Count of Participants; unit: Participants]
  Age: <5 years | 5 | 23 | 28
  Age: 5-15 years | 8 | 53 | 61
  Age: 16-44 years | 56 | 258 | 314
  Age: >45 years | 15 | 84 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 210 | 258
  Male | 36 | 208 | 244
Cycle-threshold on PCR [Median (Full Range); unit: Number of cycles] — The value represents the number of cycles the PCR has run before reaching a threshold value of a positive result.
  Number of cycles | 27.3 [19.2 to 35.8] | 26.0 [15.2 to 39.4] | 26.3 [15.2 to 39.4]
Number of participants per PCR Cycle-threshold interval [Count of Participants; unit: Participants] — The value represents the number of cycles the PCR has run before reaching a threshold value of a positive result.
  Participants
    <25 cycles | 21 | 159 | 180
    25.0-29.9 cycles | 41 | 183 | 224
    >29.9 cycles | 22 | 76 | 98
Nausea and vomiting [Count of Participants; unit: Participants] | 42 | 203 | 245
Diarrhea [Count of Participants; unit: Participants] | 29 | 155 | 184
Weakness or asthenia [Count of Participants; unit: Participants] | 77 | 353 | 430
Pain [Count of Participants; unit: Participants] | 73 | 342 | 415
Cough [Count of Participants; unit: Participants] | 11 | 40 | 51
Difficulty breathing [Count of Participants; unit: Participants] | 4 | 11 | 15
Difficulty swallowing [Count of Participants; unit: Participants] | 15 | 39 | 54
Hiccups [Count of Participants; unit: Participants] | 7 | 38 | 45
Eye redness [Count of Participants; unit: Participants] — Includes both conjunctivitis and conjunctival bleeding
  Participants | 34 | 83 | 117
Unusual bleeding [Count of Participants; unit: Participants] — Excluding conjunctival bleeding
  Participants | 5 | 21 | 26
Disorientation or agitation [Count of Participants; unit: Participants] | 0 | 2 | 2
Anuria [Count of Participants; unit: Participants] | 1 | 1 | 2
Seizures [Count of Participants; unit: Participants] | 0 | 1 | 1
Duration of symptoms >6 days [Count of Participants; unit: Participants] — Population: Only including patients with any symptom at baseline
  Participants
    number analyzed (Participants) | 73 | 412 | 485
    (all) | 14 | 203 | 217
Coexisting chronic medical condition [Count of Participants; unit: Participants]
  Infectious | 1 | 2 | 3
  Noninfectious | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Survival at Day 14 After Start of Intervention
Description: Effect of convalescent plasma in improving patients survival at day 14; it will be considered clinically significant if there is an absolute decrease in the case fatality rate of 20% or more, compared to SC alone
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard Care
Number analyzed (Participants) | 84 | 418
Participants | 58 | 260

2. Secondary Outcome: Number of Participants With 30 Days Survival
Description: Effect of convalescent plasma in improving patients survival at day 30
Time Frame: 30 days
Population: Outcome was only measured in the intervention group. Data (historical) not available for "Standard care" group.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 84
Participants | 57

3. Secondary Outcome: Titer of Ebola Viral RNA
Description: To assess the relationship between EVD antibody levels (EBOV IgG) in donated plasma and the changes in levels of viral RNA in patients who received Convalescent Plasma.
  The outcome shows the overall association between antibody dose category and change in Cycle threshold (Ct) value pre and post transfusion (Ct is the number of cycles that have to be run before reaching a threshold value of a positive result).
Time Frame: 30 days
Population: Total dose for antibody levels was categorized in three equal-sized groups (tertiles), with the lowest dose category as reference.
  71 out of 84 participants were defined as the analysis population. Children (<16 years) were excluded from the analysis as dosing of CP was done according to body weight, which was not recorded for many adult patients.
Measure: Mean (95% Confidence Interval); unit: Cycles
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 71
Cycles
  Lowest dose (antibody range 176.4 - 511.9): number analyzed (Participants) | 24
  Lowest dose (antibody range 176.4 - 511.9) | 1 [1 to 1]
  Middle dose (antibody range 513.3 - 740.6): number analyzed (Participants) | 24
  Middle dose (antibody range 513.3 - 740.6) | 3.24 [0.87 to 5.61]
  Highest dose (antibody range 747.9 - 1628.7): number analyzed (Participants) | 23
  Highest dose (antibody range 747.9 - 1628.7) | 2.34 [-0.09 to 4.78]

4. Secondary Outcome: Titer of Ebola Viral RNA
Description: To assess the relationship between EVD antibody levels (neutralizing antibodies) in donated plasma and the changes in levels of viral RNA in patients who received Convalescent Plasma.
  The outcome shows the overall association between antibody dose category and change in Cycle threshold (Ct) value pre and post transfusion (Ct is the number of cycles that have to be run before reaching a threshold value of a positive result).
Time Frame: 30 days
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Cycles
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 71
Cycles
  Lowest dose ((antibody range 176.4 - 511.9): number analyzed (Participants) | 24
  Lowest dose ((antibody range 176.4 - 511.9) | 1 [1 to 1]
  Middle dose (antibody range 513.3 - 740.6): number analyzed (Participants) | 24
  Middle dose (antibody range 513.3 - 740.6) | 0.30 [-2.30 to 2.90]
  Highest dose (antibody range 747.9 - 1628.7): number analyzed (Participants) | 23
  Highest dose (antibody range 747.9 - 1628.7) | -0.46 [-2.99 to 2.08]

5. Secondary Outcome: Number of Participants Who Died Corresponding to EV Antibody Levels (Anti-EBOV IgG)
Description: To assess the relationship between EVD antibody levels (anti-EBOV IgG) and death in patients who received Convalescent Plasma
Time Frame: 14 days
Population: Overall Number of Participants Analyzed divided in 3 equal groups depending on total dose of antibodies. 71 out of 84 participants were defined as the analysis population. Children (<16 years) were excluded from analysis as dosing of CP was done according to body weight, which was not recorded for many adult patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 71
Participants
  Low (antibody range 176.4 - 511.9): number analyzed (Participants) | 24
  Low (antibody range 176.4 - 511.9) | 5
  Medium (antibody range 513.3 - 740.6): number analyzed (Participants) | 24
  Medium (antibody range 513.3 - 740.6) | 11
  High (antibody range 747.9 - 1628.7): number analyzed (Participants) | 23
  High (antibody range 747.9 - 1628.7) | 8

6. Secondary Outcome: Number of Participants Who Died Corresponding to EV Antibody Levels (Neutralizing Antibodies)
Description: To assess the relationship between EVD antibody levels (neutralizing antibodies) and death in patients who received CP
Time Frame: 14 days
Population: Overall Number of Participants Analyzed divided in 3 equal groups depending on total dose of antibodies. Children (<16 years) were excluded from analysis as dosing of CP was done according to body weight, which was not recorded for many adult patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 71
Participants
  Low(antibody range 176.4 - 511.9): number analyzed (Participants) | 24
  Low(antibody range 176.4 - 511.9) | 6
  Medium (antibody range 513.3 - 740.6): number analyzed (Participants) | 24
  Medium (antibody range 513.3 - 740.6) | 8
  High (antibody range 747.9 - 1628.7): number analyzed (Participants) | 23
  High (antibody range 747.9 - 1628.7) | 10

7. Secondary Outcome: Number of Transfusion-related Serious Adverse Reactions (SARs)
Description: To assess the occurrence of serious adverse reactions (SARs) related to CP transfusion in Ebola patients
Time Frame: 30 days
Measure: Number; unit: SARs
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 99
SARs | 0

8. Secondary Outcome: Number of Professional Safety Incidents
Description: To assess the occurrence of safety risks related to CP transfusion in health workers administering the treatments. This will be observed throughout the study
Time Frame: 9 months
Population: Overall Number of Participants Analyzed refers to health workers administering CP; not to the participants receiving CP.
Measure: Number; unit: Professional safety incidents
Arm/Group | Convalescent Plasma
Number analyzed (Participants) | 12
Professional safety incidents | 0

9. Secondary Outcome: Mortality Risk Factor: Ct
Description: To determine Ct as risk factor for mortality despite administration of CP.
Time Frame: 30 days
Population: Pre-specified sub-group comparison
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard Care
Number analyzed (Participants) | 84 | 418
Participants
  10-24.9 cycles: number analyzed (Participants) | 21 | 159
  10-24.9 cycles | 11 | 90
  25-29.9 cycles: number analyzed (Participants) | 41 | 183
  25-29.9 cycles | 11 | 56
  30-39.9 cycles: number analyzed (Participants) | 22 | 76
  30-39.9 cycles | 4 | 12

10. Secondary Outcome: Mortality Risk Factor: Age
Description: To determine age as risk factor for mortality despite administration of CP.
Time Frame: 30 days
Population: Pre-specified sub-group comparison
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard Care
Number analyzed (Participants) | 84 | 418
Participants
  <5 years old: number analyzed (Participants) | 5 | 23
  <5 years old | 1 | 15
  5-15 years old: number analyzed (Participants) | 8 | 53
  5-15 years old | 1 | 10
  16-44 years old: number analyzed (Participants) | 56 | 258
  16-44 years old | 16 | 90
  >45 years old: number analyzed (Participants) | 15 | 84
  >45 years old | 8 | 43

ADVERSE EVENTS:
Time Frame: All adverse events related to the intervention up to 4 hours after completion of the transfusion. All deaths possibly related to the intervention up to 14 days after completion of the transfusion.
Description: Due to the nature of the symptoms of EVD (high mortality rate, hospital admissions, disability and life-threatening conditions), the investigation of safety and tolerability of the intervention will focus on Adverse Reactions.
  An Adverse Reaction is any untoward and unintended response in a participant to the study treatment, which is related (or has a reasonable possibility of being related) to any dose of the investigational product administered to that participant.
Groups:
- Convalescent Plasma: Convalescent Plasma: 400-500 mL from two donors (2 x 200-250 ml) and 10mL/kg for small adults and children <45kg
  Convalescent Plasma: Patients will be treated with plasma from recovered EVD patients.
  No data from "standard care" group available as this is based on historical data.
Arm/Group | Convalescent Plasma
All-Cause Mortality (participants affected / at risk) | 26/84
Serious Adverse Events (participants affected / at risk) | 0/84
Other Adverse Events (participants affected / at risk) | 8/84
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Plasma (N=84)
Increase in temperature (General disorders) | 5
Itching or skin rash (Skin and subcutaneous tissue disorders) | 4
Nausea (General disorders) | 1

LIMITATIONS AND CAVEATS:
There are clear limitations with respect to the use of a historical control group, and we cannot exclude the possibility that unmeasured confounding factors may have biased the mortality comparison.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes